CLINICAL TRIAL: NCT02398552
Title: A Randomized Phase II Trila of Sunitinib Four-weeks on/Two-weeks Off Versus Two-weeks on/One-week Off as First Line Therapy in Metastatic Renal Cell Carcinoma.
Brief Title: A Phase II Trila of Sunitinib Schedule 4/2 vs. Shedule 2/1 as First Line Therapy in Metastatic Renal Cell Carcinoma.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun Guo, Director of department of renal cancer and melanoma, Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCH-RCC-150212
Record Dates: First submitted 2015-03-20; First posted 2015-03-25 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: metastatic renal cell carcinoma; sunitinib; schedule 2weeks on/1 week off
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sunitinib 50mg/day schedule 4/2 (Active Comparator): Sunitinib 50mg/day 4 weeks on/2 weeks off per 6 weeks till disease progression or intolerable toxicity.
  Interventions: Drug: Sunitinib
- Sunitinib 50mg/day schedule 2/1 (Experimental): Sunitinib 50mg/day 2 weeks on/1 week off per 6 weeks till disease progression or intolerable toxicity.
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — altenative schedules of sunitinib as first line therapy in metastatic renal cell carcinoma patients.
  Other Names: Sutent

SUMMARY:
Sunitinib given at 50 mg/day on schedule 4/2 (4 weeks on treatment, 2 weeks off) is the standard care for first-line treatment of metastatic renal cell carcinoma, but the schedule was reported with a high rate of dose reduction and dose discontinuation because of the safety profile. So investigators conducte this randomized, multi-center phase II study to determine whether a sunitinib regimen of 50 mg/day 2-weeks on/1-week off could provide the same efficacy in terms of progression-free survival, objective response, and overall survival, while reducing drug-related toxicity.

DETAILED DESCRIPTION:
Sunitinib given at 50 mg/day on schedule 4/2 (4 weeks on treatment, 2 weeks off) is the standard care for first-line treatment of metastatic renal cell carcinoma, but the schedule was reported with a high rate of dose reduction and dose discontinuation because of the safety profile. Sunitinib 50mg/day on schedule 2/1 (2 weeks on treatment, 1 weeks off) was reported to be associated with significantly decrease toxicities in patients who initially experienced grade 3 or greater toxicity on the schedule 4/2 and could extend treatment duration considerably. Through this research, we would like to explore whether the schedule 2/1 of sunitinib 50 mg/day as first line therapy could provide the same efficacy as standard schedule 4/2 in terms of progression-free survival, objective response, and overall survival, while reducing drug-related toxicity in metastatic renal cell carcinoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years, ≤75 years, male or female
* Advanced renal cell carcinoma is diagnosed histologically or pathologically
* Treatment naive at diagnosed
* At least one measurable tumor lesion (Response Evaluation Criteria In Solid Tumors)
* Eastern Cooperative Oncology Group（ECOG) performance scale is 0 or 1
* The expected life span is ≥12 weeks
* No contraindications for targeted therapy, with enough liver function and renal function and normal ECG recording Peripheral hemogram: neutrophil≥1.5×109/L, Plt≥100×109/L, Hgb≥90g/L Renal function: serum creatinine≤1.5 folds the upper limit of normal (ULN) For patients with non-metastatic liver dysfunction:alanine aminotransferase and aspartate aminotransferase≤2.5 ULN, For patients with metastatic liver dysfunction: alanine aminotransferase and aspartate aminotransferase≤5 ULN
* The patients participate voluntarily and have signed the informed consent form

Exclusion Criteria:

* Patients who have received any systemic therapy including targeted therapy,immunotherapy,chemotherapy etc at diagnosed.
* Pregnant and lactating women, or female patients of child-bearing age without taking contraceptive measures
* Patients with severe acute infection without being controlled effectively or having pyogenic and chronic infections with persistently unhealed wounds
* Past history of serious heart diseases, including: cardiac function classification ≥NYHA class II, unstable angina pectoris, myocardial infarction, arrhythmia requiring anti-arrhythmic drug therapy (excluding β-blockers or digoxin), and uncontrolled hypertension
* Patients with a history of HIV infection or active phase of chronic hepatitis B/C
* negative imaging examination result 4 weeks prior to enrollment)
* Epilepsy patients requiring drug therapy (e.g. steroids or antiepileptic drugs)
* A history of allogeneic organ transplantation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
progress-free survival (PFS) | 2 years
  Time from enrollment to the dates of disease progression,death from any cause or last tumor assessment reported between date of first patient enrollment until March 2017 cut off date

SECONDARY OUTCOMES:
The percentage of patients who can get complete response, partial response. | 2 years

OTHER OUTCOMES:
Number of adverse events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, MD,PHD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (6):
- China (6):
  - Chinese acadamy of medical science cancer institute & hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen university cancer center, Guangzhou, Guangdong
  - Cancer Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Tianjin medical university cancer institute & hospital, Tianjin, Tianjin Municipality

REFERENCES:
- [Background] Motzer RJ, Hutson TE, Tomczak P, Michaelson MD, Bukowski RM, Oudard S, Negrier S, Szczylik C, Pili R, Bjarnason GA, Garcia-del-Muro X, Sosman JA, Solska E, Wilding G, Thompson JA, Kim ST, Chen I, Huang X, Figlin RA. Overall survival and updated results for sunitinib compared with interferon alfa in patients with metastatic renal cell carcinoma. J Clin Oncol. 2009 Aug 1;27(22):3584-90. doi: 10.1200/JCO.2008.20.1293. Epub 2009 Jun 1. PMID 19487381
- [Background] Houk BE, Bello CL, Poland B, Rosen LS, Demetri GD, Motzer RJ. Relationship between exposure to sunitinib and efficacy and tolerability endpoints in patients with cancer: results of a pharmacokinetic/pharmacodynamic meta-analysis. Cancer Chemother Pharmacol. 2010 Jul;66(2):357-71. doi: 10.1007/s00280-009-1170-y. Epub 2009 Dec 5. PMID 19967539
- [Background] Neri B, Vannini A, Brugia M, Muto A, Rangan S, Rediti M, Tassi R, Cerullo C. Biweekly sunitinib regimen reduces toxicity and retains efficacy in metastatic renal cell carcinoma: a single-center experience with 31 patients. Int J Urol. 2013 May;20(5):478-83. doi: 10.1111/j.1442-2042.2012.03204.x. Epub 2012 Nov 1. PMID 23113655